CLINICAL TRIAL: NCT03787927
Title: Reversal of Dual Antiplatelet Therapy With Cold Stored Platelets
Acronym: R-DAPT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bloodworks (Other)
Collaborators: National Blood Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-02
Record Dates: First submitted 2018-12-19; First posted 2018-12-27 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Bleeding; Platelet Dysfunction Due to Drugs; Platelet Dysfunction
MeSH Terms: conditions — Hemorrhage | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 5 day CSP, then 5 day RTP (Other): Participants will first complete collection and transfusion of 5 day autologous CSP (cold-stored platelet). Then they will complete collection and transfusion of 5 day autologous RTP (room-temperature-stored platelets). The day before each transfusion, Aspirin (325mg) and Clopidogrel (600mg) will be administered.
  The first 20 participants who complete the study will be randomized to this arm or '5 day RTP, then 5 day CSP.'
  Interventions include: Aspirin, Clopidogrel, Autologous Platelet Transfusion (cold-stored 5 days), Autologous Platelet Transfusion (room-temperature-stored 5 days)
  Interventions: Drug: Autologous Platelet Transfusion (room-temperature-stored); Drug: Autologous Platelet Transfusion (cold-stored 5 days); Drug: Aspirin; Drug: Clopidogrel
- 5 day RTP, then 5 day CSP (Other): Participants will first complete collection and transfusion of 5 day autologous RTP (room-temperature-stored platelets). Then they will complete collection and transfusion of 5 day autologous CSP (cold-stored platelets). The day before each transfusion, Aspirin (325mg) and Clopidogrel (600mg) will be administered.
  The first 20 participants who complete the study will be randomized to this arm or '5 day CSP, then 5 day RTP.'
  Interventions include: Aspirin, Clopidogrel, Autologous Platelet Transfusion (cold-stored 5 days), Autologous Platelet Transfusion (room-temperature-stored 5 days)
  Interventions: Drug: Autologous Platelet Transfusion (room-temperature-stored); Drug: Autologous Platelet Transfusion (cold-stored 5 days); Drug: Aspirin; Drug: Clopidogrel
- 5 day RTP, then 10 day CSP (Other): Participants will first complete collection and transfusion of 5 day autologous RTP (room-temperature-stored platelets). Then they will complete collection and transfusion of 10 day autologous CSP (cold-stored platelets).The day before each transfusion, Aspirin (325mg) and Clopidogrel (600mg) will be administered.
  After the first 20 complete data sets are obtained from subjects, the next 20 complete data sets will be obtained (if progression to this arm is indicated) by randomizing subjects between '5 day RTP, then 10 day CSP' and '10 day CSP, then 5 day RSP.'
  Interventions include: Aspirin, Clopidogrel, Autologous Platelet Transfusion (cold-stored 10 days), Autologous Platelet Transfusion (room-temperature-stored 5 days)
  Interventions: Drug: Autologous Platelet Transfusion (room-temperature-stored); Drug: Autologous Platelet Transfusion (cold-stored 10 days); Drug: Aspirin; Drug: Clopidogrel
- 5 day RTP, then 15 day CSP (Other): Participants will first complete collection and transfusion of 5 day autologous RTP (room-temperature-stored platelets). Then they will complete collection and transfusion of 15 day autologous CSP (cold-stored platelets). The day before each transfusion, Aspirin (325mg) and Clopidogrel (600mg) will be administered.
  After the first 40 complete data sets are obtained from subjects, the next 20 complete data sets will be obtained (if progression to this arm is indicated) by randomizing subjects between '5 day RTP, then 15 day CSP' and '15 day CSP, then 5 day RSP.'
  Interventions include: Aspirin, Clopidogrel, Autologous Platelet Transfusion (cold-stored 15 days), Autologous Platelet Transfusion (room-temperature-stored 5 days)
  Interventions: Drug: Autologous Platelet Transfusion (room-temperature-stored); Drug: Autologous Platelet Transfusion (cold-stored 15 days); Drug: Aspirin; Drug: Clopidogrel
- 10 day CSP, then 5 day RTP (Other): Participants will first complete collection and transfusion of 10 day autologous CSP (cold-stored platelet). Then they will complete collection and transfusion of 5 day autologous RTP (room-temperature-stored platelets).The day before each transfusion, Aspirin (325mg) and Clopidogrel (600mg) will be administered.
  After the first 20 complete data sets are obtained from subjects, the next 20 complete data sets will be obtained (if progression to this arm is indicated) by randomizing subjects between '5 day RTP, then 10 day CSP' and '10 day CSP, then 5 day RSP.'
  Interventions include: Aspirin, Clopidogrel, Autologous Platelet Transfusion (cold-stored 10 days), Autologous Platelet Transfusion (room-temperature-stored 5 days)
  Interventions: Drug: Autologous Platelet Transfusion (room-temperature-stored); Drug: Autologous Platelet Transfusion (cold-stored 10 days); Drug: Aspirin; Drug: Clopidogrel
- 15 day CSP, then 5 day RTP (Other): Participants will first complete collection and transfusion of 15 day autologous CSP (cold-stored platelet). Then they will complete collection and transfusion of 5 day autologous RTP (room-temperature-stored platelets). The day before each transfusion, Aspirin (325mg) and Clopidogrel (600mg) will be administered.
  After the first 40 complete data sets are obtained from subjects, the next 20 complete data sets will be obtained (if progression to this arm is indicated) by randomizing subjects between '5 day RTP, then 15 day CSP' and '15 day CSP, then 5 day RSP.'
  Interventions include: Aspirin, Clopidogrel, Autologous Platelet Transfusion (cold-stored 15 days), Autologous Platelet Transfusion (room-temperature-stored 5 days)
  Interventions: Drug: Autologous Platelet Transfusion (room-temperature-stored); Drug: Autologous Platelet Transfusion (cold-stored 15 days); Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Autologous Platelet Transfusion (room-temperature-stored) — The participant will receive an autologous platelet transfusion of their room-temperature-stored platelets after 5 days of storage.
Drug: Autologous Platelet Transfusion (cold-stored 5 days) — The participant will receive an autologous platelet transfusion of their cold-stored platelets after 5 days of storage.
  Arms: 5 day CSP, then 5 day RTP; 5 day RTP, then 5 day CSP
Drug: Autologous Platelet Transfusion (cold-stored 10 days) — The participant will receive an autologous platelet transfusion of their cold-stored platelets after 10 days of storage.
  Arms: 10 day CSP, then 5 day RTP; 5 day RTP, then 10 day CSP
Drug: Autologous Platelet Transfusion (cold-stored 15 days) — The participant will receive an autologous platelet transfusion of their cold-stored platelets after 15 days of storage.
  Arms: 15 day CSP, then 5 day RTP; 5 day RTP, then 15 day CSP
Drug: Aspirin — Aspirin (325mg) will be administered the day before every transfusion.
Drug: Clopidogrel — Clopidogrel (600mg) will be administered the day before every transfusion.

SUMMARY:
This study aims to determine whether cold-stored platelets (CSP) are equally, more effective, or uniquely effective at reversing the effect of dual antiplatelet therapy in healthy human subjects compared to room-temperature-stored platelets (RTP). The investigators plan to enroll healthy human subjects without risk factors for bleeding to achieve 60 complete data sets. Each subject will donate two apheresis platelet units. One platelet unit will be stored in the cold (CSP) and one platelet unit will be stored at room temperature (RTP). Subjects will be given dual anti-platelet therapy (aspirin and clopidogrel) prior to autologous transfusion of each unit. Platelet function testing will be performed before and after transfusion to measure reversal of the antiplatelet drugs.

ELIGIBILITY:
Inclusion Criteria:

The subject is in good health, is taking no excluded medications and meets platelet donor suitability requirements aimed at assuring donor safety.

1. Subject self-reports that he or she feels well and healthy
2. Subjects must be 18-59 years old, of either sex
3. Temperature: less than or equal to 99.5 F
4. Resting blood pressure: systolic less than or equal to 180 mmHg, diastolic less than or equal to100 mmHg
5. Resting heart rate: 40 to 100 beats per minute
6. Weight: greater than or equal to110 pounds,
7. Hematocrit: greater than or equal to 35 percent for females, greater than or equal to 38 percent for males, but not greater than 55 percent
8. Platelet count able to achieve target platelet yield per apheresis machine configuration parameters
9. Subjects must be able to read, understand and sign the informed consent document and commit to the study follow-up schedule. The ability to read and speak English is required for participation.
10. Subject must agree to avoid taking any aspirin or aspirin-containing drugs (e.g., Alka-Seltzer, Bufferin, Excedrin) or NSAIDs (e.g.,Feldene, Motrin, Aleve, Advil) or other drugs known to affect platelet function throughout their study participation.
11. Subjects must agree to avoid calcium channel blockers such as amlodipine (Norvasc), felodipine, and verapamil (Verelan, Calan) and proton pump inhibitors (PPIs) such as omeprazole (Prilosec), lansoprazole (Prevacid), esomeprazole (Nexium) and pantoprazole (Protonix) until all study blood draws are concluded. These classes of drugs may interfere with the action of clopidogrel and diminish its antiplatelet effect.
12. Subjects must have "good veins" for apheresis platelet collection and drawing blood samples.
13. Women of child bearing potential must agree to use an effective method of contraception during the course of the study. The following methods of contraception will be considered 'effective' when self-reported by subject; abstinence, intrauterine contraception devices, hormonal methods, barrier methods or history of sterilization.
14. Subject has phone and e-mail for contact and notification, and is able to come to the research site for approximately 9 visits over up to approximately 64 days.

Exclusion Criteria:

Healthy subjects will be excluded from the study for any of the following reasons:

1. Active acute infection or suspected active infection, temperature above 100 F or taking antibiotic
2. Active immune/inflammatory condition (e.g. gout, systemic lupus erythematosus, allograft rejection)
3. History of heart disease, including endorsement of shortness of breath with mild exertion (at the discretion of the PI).
4. History of significant liver, kidney, GI, blood, endocrine/metabolic, autoimmune or pulmonary disease, untreated hypertension and or metabolic syndrome (at the discretion of the PI).
5. Diabetes Mellitus
6. Cancer of any kind (exceptions being basal or squamous cell cancers of the skin), under treatment or resolved
7. History of bleeding events, family history of bleeding events, or known genetic disorder with bleeding diathesis
8. A family history of venous or arterial thrombosis before the age of 50 in first degree relatives
9. A personal history of DVT, venous or arterial thrombosis, blood clots or stroke
10. History of having been prescribed clopidogrel (Plavix), ticlopidine (Ticlid) or Ticagrelor (Brilinta).
11. Subject has taken any aspirin or aspirin-containing drugs (e.g., Alka-Seltzer, Bufferin, Excedrin) or NSAIDs (e.g.,Feldene, Motrin, Aleve, Advil) or other drugs known to affect platelet function within 14 days prior to screening.
12. Chronic NSAID therapy
13. Chronic steroid therapy
14. Known allergy to aspirin or clopidogrel
15. Subjects who are taking, or have taken within 14 days any of the following class of drugs protone pump inhibitors (PPIs) such as omeprazole, pantoprazole, lansoprazole, esomeprazole lipid lowering drugs/statins anticoagulants ACE-inhibitors phenytoine tolbutamide calcium channel blockers such as amlodipine, felodipine, verapamil
16. Current drug or alcohol dependence by subject's declaration.
17. Currently pregnant or nursing as assessed during interview. A urine pregnancy test prior to apheresis is required for women of childbearing potential.
18. Subject plans to participate in contact sports during study/observational period such as boxing, rugby, American football, soccer, or other risky recreational hobbies at the discretion of the investigator.
19. Unwilling or unable to comply with the protocol in the opinion of the investigator.
20. Participation in an experimental drug/device study within the past 30 days (other than this study). Subjects who have received an infusion on this study may not be re-enrolled.
21. Average initial (only for the first PFT) aggregation responses to ADP less than or equal to 60% by aggregometry platelet function testing.
22. Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-12-03 (Estimated); Study Completion 2021-12-03 (Estimated)

PRIMARY OUTCOMES:
Verify Now (PRU): αIIbβ3 (GPIIb-IIIa) integrin activation changes between DAPT loaded pre-transfusion, 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion, baseline | Measured at baseline, pre-transfusion (after administration of dual anti-platelet therapy), 1 hour post-transfusion, 24 hour post-transfusion
  Measured by Verify Now (PRU)
Verify Now: αIIbβ3 (GPIIb-IIIa) integrin activation changes between DAPT loaded pre-transfusion, 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion, baseline | Measured at baseline, pre-transfusion (after administration of dual anti-platelet therapy), 1 hour post-transfusion, 24 hour post-transfusion
  Measured by Verify Now (ARU)
PAC-1: αIIbβ3 (GPIIb-IIIa) integrin activation changes between DAPT loaded pre-transfusion, 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion, baseline | Measured at baseline, pre-transfusion (after administration of dual anti-platelet therapy), 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion
  Measured by PAC-1 antibody binding by flow cytometry

SECONDARY OUTCOMES:
LTA: αIIbβ3 (GPIIb-IIIa) integrin activation changes from DAPT loaded pre-transfusion, 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion, baseline | Measured at baseline, pre-transfusion (after administration of dual anti-platelet therapy), 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion
  Light Transmittance Aggregometry
P-Selectin:αIIbβ3 (GPIIb-IIIa) integrin activation changes between DAPT loaded pre-transfusion, 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion, baseline | Measured at baseline, pre-transfusion (after administration of dual anti-platelet therapy), 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion
  Measured by alpha-granule secretion (P-Selectin) by flow cytometry
Beeding time testing (in-vivo) changes between DAPT loaded pre-transfusion, 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion, baseline | Measured at baseline, pre-transfusion (after administration of dual anti-platelet therapy), 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion
  in-vivo subject testing
CBC changes between DAPT loaded pre-transfusion, 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion, baseline | Measured at baseline, pre-transfusion (after administration of dual anti-platelet therapy), 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion
Platelet unit blood gas: changes during storage | day of collection, day of transfusion
  during storage of the units
Platelet unit Annexin V: changes during storage | day of collection, day of transfusion
Thromboxane B2 ELISA changes between DAPT loaded pre-transfusion, 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion, baseline | Measured at baseline, pre-transfusion (after administration of dual anti-platelet therapy), 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion
Vasodilator-stimulated phosphoprotein (VASP) changes | Measured at baseline, pre-transfusion (after administration of dual anti-platelet therapy), 1 hour post-transfusion, 4 hour post-transfusion, 24 hour post-transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Stolla, MD, Principal Investigator — Bloodworks Northwest
Locations (1):
- Bloodworks Northwest Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miles J, Bailey SL, Obenaus AM, Mollica MY, Usaneerungrueng C, Byrne D, Fang L, Flynn JR, Corson J, Osborne B, Houck K, Wang Y, Shen Y, Fu X, Dong JF, Sniadecki NJ, Stolla M. Storage temperature determines platelet GPVI levels and function in mice and humans. Blood Adv. 2021 Oct 12;5(19):3839-3849. doi: 10.1182/bloodadvances.2021004692. PMID 34478498